CLINICAL TRIAL: NCT06039956
Title: De-escalating Axillary Surgery After Neoadjuvant Chemotherapy in Node Positive Breast Cancer Patients in Nigeria
Brief Title: De-escalating Axillary Surgery in Breast Cancer Patients in Nigeria
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Obafemi Awolowo University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0004553
Record Dates: First submitted 2023-04-11; First posted 2023-09-15 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Axilla; Breast
Keywords: neoadjuvant; de-escalation; breast cancer; axillary lymph node staging
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel Lymph Node Biopsy Arm (Other): Patients with non-metastatic, biopsy and clipped locally advanced breast cancer will start systemic chemotherapy as per institutional best practices. Patients with a clinical complete response will be consented for SLNB followed by immediate ALND. Patients with persistent suspicious clinical adenopathy will be consented for ALND alone. All patients regardless of response to NAC will undergo ALND as per current institutional practices.
  Patients undergoing SLNB followed by ALND will have the procedure performed by study the co-PI at OAUTH who is trained in the performance of SLNB. Histopathologic assessment of the breast and axillary contents will follow a standardized reporting procedure, including the assessment of residual cancer burden in both the breast and the axilla. Presence or absence of residual disease will be reported separately for the SLNB specimens, clipped node and remaining axillary contents.
  Interventions: Procedure: Sentinel lymph Node Biopsy

INTERVENTIONS:
Procedure: Sentinel lymph Node Biopsy — The SLNB will be performed with 5 ml of undiluted methylene blue injected in equal aliquots, peri-tumoral, followed by a 5-minute massage prior to skin incision. Sentinel nodes will be defined as those that have uptake / visible blue staining or suspicious palpable nodes at the discretion of the operating surgeon. Sentinel nodes will be placed in formalin and sent separately. This will be followed by an immediate completion ALND, which will be similarly placed in formalin and sent separately from the SLNB specimen. Specimen radiographs will be performed on all specimens to confirm location of clip within SLNB vs. ALND specimens.

SUMMARY:
In sub-Saharan Africa, breast cancer patients often present with advanced disease. In my previous research which evaluated over 600 patients from a prospective institutional data base, about 64% of women with a new diagnosis of breast cancer presented with locally advanced disease, including clinically positive axillary adenopathy. Our data also suggests that similar to African American women, triple negative breast cancer (TNBC) is common in Nigeria (43.5%).

The overall goal of the project is to evaluate the ability of existing technology in Nigeria to safely de-escalate axillary surgery in the management of locally advanced breast cancer patients. Currently, the standard-of-care for breast cancer patients with palpable axillary adenopathy (clinical N1 disease without evidence of distant metastases) at presentation in Nigeria is neoadjuvant systemic therapy followed by a modified radical mastectomy. This includes a complete axillary lymph node dissection (ALND). However, data from high-income countries however show that up to 85% of patients initially presenting with cN1 disease can be converted to cN0 (i.e. no palpable adenopathy) following NAC. These patients can thus safely undergo sentinel lymph node biopsy (SLNB) with up to 50% of these having pathologic complete response in the lymph nodes. In this patient population, both methylene blue and radio-isotope localization with Tc-99 sulphur colloid are required to ensure adequate performance of the SLNB to stage the axilla(i.e. false negative rate ≤10%). Although widely available in high-income countries, radio-isotope localization is not readily available in Nigeria. This project will explore an alternative to dual agent SLNB localization using readily available resources and multi-disciplinary collaboration in a lower-income environment. De-escalation of axillary surgery in high-income countries has significantly decreased operative morbidity and improved patient reported outcomes without compromising survival. However, context specific research and data from resource limited environments is needed to translate the benefit of de-escalation to sub-Saharan Africa.

DETAILED DESCRIPTION:
The overall goal of my research is to promote the delivery of guideline-concordant breast cancer care to Nigerian breast cancer patients in a pragmatic manner. This project is novel in that the investigators are challenging the existing paradigm of dual agent localization, which is appropriate for a high-income setting, but completely out of reach and thus inapplicable in Nigeria despite the obvious need. I will leverage the African Research Group for Oncology (ARGO) breast cancer data base at OAUTHC and other existing research infrastructure to pursue the following specific aims: Aim 1: Determine the false negative rate of of axillary Ultrasound + single agent sentinel Lymph node biopsy in staging the axilla in cN1 patients who become cN0. The investigators will consent patients with complete clinical complete response (clinical assessment and targeted US) following NAC, for SLNB followed by immediate ALND. Presence or absence of residual disease will be reported separately for the SLNB and the ALND specimens. Positive axillary disease will be defined in a binary manner as any invasive disease (including isolated tumor cells) or not. Using ALND reporting as the gold standard, the investigators hypothesize a FNR of less than 10% following SLNB. Aim 2: To determine the proportion of patients with complete axillary LN Clinical &Pathological cR post NAC. The proportion of patients who return negative for cancer cells following SLNB and or ALND will be determined based on the number of patients with preoperative node positive disease. Both overall pCR and subgroup analysis based on receptor status will be done. The investigators will also assess the concordance of pre-operative clinical and radiographic (i.e. targeted axillary US) assessment of lymph node status with and pathologic lymph node status after NAC. The investigators hypothesize a pCR rate of 50% following completion of NAC

This study will build on the peer-reviewed analysis of our own prospective data demonstrating a high incidence of locally advanced disease and chemo-sensitive subtypes (i.e. TNBC), which suggest that a large proportion of our patients may be candidates for de-escalation. The impact of de-escalation would be profound. Preliminary research into lymphedema as a result of ALND in our patient population suggest an incidence of > 35%. The proposed study will provide a strong foundation for future studies evaluating the implementation of this strategy and other resource compatible interventions on breast cancer outcomes in Nigeria.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to receive systemic chemotherapy

Must include all the following:

* Tany, cN1 at presentation
* Biopsy proven pN1 disease after axillary US
* cN0 after neoadjuvant chemotherapy

Exclusion Criteria:

* Previous / recurrent breast cancer
* Previous axillary and/or breast surgery
* Inflammatory breast cancer
* N2 disease or Stage IV disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
False-negative rate | immediately after surgery
  • False negative rate (FNR) of pre-op axillary US and single agent SLNB post-NAC for axillary staging

SECONDARY OUTCOMES:
pathologic complete response rate | immediately after surgery
  • Incidence of axillary lymph node clinical and pathologic complete response in patient receiving NAC in Nigeria
radiographic and clinical concordance | immediately after surgery
  • Concordance of pre-operative clinical, radiographic and pathologic lymph node status after NAC
Sensitivity of pre-operative axillary US | immediately after surgery
  • Performance of pre-operative axillary US to stage the axilla in node positive patients who are cN0 disease after NAC
Specificity of pre-operative axillary US | immediately after surgery
  • Performance of pre-operative axillary US to stage the axilla in node positive patients who are cN0 disease after NAC
False negative rate of pre-operative axillary US | immediately after surgery
  • Performance of pre-operative axillary US to stage the axilla in node positive patients who are cN0 disease after NAC
Sensitivity of single-agent sentinel lymph node biopsy | immediately after surgery
  • Performance of single agent SLNB using methylene blue to stage the axilla in node positive patients who are cN0 disease after NAC
Specificity of single-agent sentinel lymph node biopsy | immediately after surgery
  • Performance of single agent SLNB using methylene blue to stage the axilla in node positive patients who are cN0 disease after NAC
False negative rate of single-agent sentinel lymph node biopsy | immediately after surgery
  • Performance of single agent SLNB using methylene blue to stage the axilla in node positive patients who are cN0 disease after NAC

CONTACTS AND LOCATIONS:
Overall Officials: Olalekan Olasenhinde, MD, Principal Investigator — Obafemi Awolowo University